CLINICAL TRIAL: NCT04588870
Title: Pilot Clinical Study Using Pre-operative Simulation for Patients Undergoing Cochlear Implant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was never funded.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other); Region Capital Denmark (Other)
Responsible Party: Principal Investigator, Gregory Wiet, Professor of Otolaryngology, Pediatrics and Biomedical Informatics, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OSU2020H0080
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Sensori-Neural Deafness
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Cochlear Implant (Experimental): The intervention will be the use of a surgical simulation system preoperatively by the surgeon to develop the surgical plan to optimize electrode array placement with respect to scalar location and modiolar distance.
  Interventions: Device: Pre operative computer based cochlear implant surgical simulation

INTERVENTIONS:
Device: Pre operative computer based cochlear implant surgical simulation — Prior to surgery, the surgeon will perform virtual cochlear implant surgery on patient specific imaging data within a computer simulation program. The surgeon will be able to iterate the procedure on the simulator until achieving the best electrode array location is achieved with respect to scalar location and modiolar distance. A written and graphical surgical plan will then be developed that the surgeon can use in the actual surgery.

SUMMARY:
36 patients will be enrolled in a pilot trial. Eligible patients (receiving CI at OSU) that consent to participate into the study will be enrolled. A simulation with visualize cochlear substructures will be created for each patient, and surgeon will conduct virtual surgery with various cochlear implant electrode types and using different techniques for optimal positioning. Based on the feedback from the simulation platform, the surgeon will find the optimal CI electrode and surgical technique using the virtual simulation and a formal plan will be recorded to guide the actual surgery. Patient demographic information, medical history and pre op audiogram will be collected once enrolled. Post-op images will be used to identify the actual electrode location (scalar location (SL), modiolar distance (MD) and and angular insertion depth (AID). At 6- and 12-months post-op, word score (CNC) will be obtained as primary clinical outcomes and AZBio scores will also be obtained and evaluated as a secondary clinical outcome. All outcomes data to be collected for SA3 are considered as part of routine clinical care for patients undergoing CI at our institution. The prospective data collection plan will ensure these data will be collected timely with high quality. OSU IRB approval has been obtained for this study (OSU IRB# 2020H0080: Virtual Reality simulation for patient specific surgical rehearsal in cochlear implantation - OSU#2) pending additional amendments as needed.

DETAILED DESCRIPTION:
Hypothesis: Patients undergoing pre-operative CI simulation will have improved outcomes as measured by SL, MD and audiological outcomes.

The goal of this aim is to demonstrate clinical feasibility and to collect preliminary efficacy data for using the pre-operative simulation with active feedback for CI patients. This will be achieved by prospectively using the CI simulation system and evaluating both technical and clinical audiological outcomes.

C.4.1 Pre-operative Simulation: Prior to surgery, a simulation with visualization of cochlear microstructures will be created for each patient, and the surgeon will conduct iterative virtual surgery with active feedback to determine the optimal surgical approach and cochlear implant electrode position. Based on the feedback from the simulation platform, the surgeon will determine the optimal CI electrode and surgical technique using the virtual simulation to plan the actual surgery. Post-implant feedback will be displayed to the surgeon. Once parameters (SL, MD, AID) are optimized, a surgical plan will be recorded and used during the actual surgical procedure. A surgical plan will consist of the implant type, cochleostomy site, and insertion techniques used for optimal placement. This will be added to the patient electronic medical record to be referenced immediately prior to surgery. Additionally, the simulator will save all performances with the optimized performance being made available for review on the simulator at any time (3-dimensional playback).

C.4.2 Clinical Outcomes: Aided speech perception testing in the CI ear will be administered at 6- and 12-months post activation using monosyllabic words (CNC Word test) presented at 60 dB SPL (A-weighted) as well as sentences (AzBio) in quiet and at +10 signal-to-noise ratio. Percent correct will be calculated for each test and will serve as the primary clinical outcomes.

C.4.3 User Evaluation: Simulator evaluation (user interface, usefulness, potential usage in future, and overall satisfactory) and feedback/comments from the surgeon about the simulation platform will continued to be collected pre and post-operatively to provide insight into continued future improvement of the simulation platform.

C.4.5 Reproducibility and Rigor:

Statistical Analysis: Demographic information as well as post-op CI location parameters (SL, MD, AID), pre/post-op CNC and AzBio scores will be summarized with descriptive statistics: mean/SD, median/IQR for continuous variables and count/percentage for categorical data. Changes of the CNC /AzBio scores overtime will be analyzed using linear mixed models to account for the association of measures from the same patient at different time points, and to deal with missing data assuming missing data will occur randomly. Exploratory analysis will be conducted to (1) evaluate the association of the CI location parameters with the post-op CNC scores; (2) compare the post-op CI location parameters with the CI patients without pre-op simulations that are reported in the literature and/or those who have undergone CI insertion in this institution (historical controls at OSU).

Sample Size: For this pilot study, a sample size of 30 patients is proposed to evaluate selected feasibility issues, assess the adequacy of instrumentation, and collect preliminary efficacy data (along with historical data) for the design of a larger prospective, randomized trial. For the improvement of the clinical outcome (CNC) after CI, a sample size of 30 patients produces a one-sided 90% upper confidence limit of variance <1.5 when the sample variance of the improvement of CNC is 1.0. Up to 36 patients will be enrolled to account for potential attrition due to various unexpected reasons during the period from the enrollment to implant surgery, to 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural Deafness
* Candidate for cochlear implantation

Exclusion Criteria:

* Inability to participate
* Not a candidate for cochlear implantation
* Age less than 18 or greater than 90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change of CNC score | 6 months after cochlear implantation compared to pre surgery.
  Aided speech perception testing in the CI ear, higher percent score (up to 100) means better hearing outcome. Range is from 0 to 100%.

SECONDARY OUTCOMES:
AZBio scores | 6 months after cochlear implantation
  Aided speech perception testing in the CI ear, higher percent score (up to 100) means better hearing outcome. Range is from 0 to 100%.
CNC scores | 12 months after cochlear implantation
  Aided speech perception testing in the CI ear, higher percent score (up to 100) means better hearing outcome. Range is from 0 to 100%.
AZBio scores | 12 months after cochlear implantation
  Aided speech perception testing in the CI ear, higher percent score (up to 100) means better hearing outcome. Range is from 0 to 100%.

OTHER OUTCOMES:
Scalar Location | 1 to 4 weeks after surgery (first post op imaging)
  location of the electrode array within the cochlear with respect to scalar
Modiolar Distance | 1 to 4 weeks after surgery (first post op imaging)
  electrode distance from the mid-modiolar line as an approximation of the distance to the spiral ganglion nerves.

IPD SHARING:
Plan to Share IPD: No